CLINICAL TRIAL: NCT04571255
Title: Music Therapy and Pain Management in Burn Patients At the Adults Intensive Care Unit of the University Hospital Fundación Santa Fe De Bogotá, Colombia.
Brief Title: Music Therapy and Pain Management in Burn Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Collaborators: University of Los Andes, Columbia (Other)
Responsible Party: Principal Investigator, Mark Ettenberger, Coordinator Music Therapy, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTUCIA01
Record Dates: First submitted 2020-05-29; First posted 2020-09-30 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Burns; Pain
Keywords: music therapy; burn patients; intensive care; pain
MeSH Terms: conditions — Burns; Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive a minimum of 3 and a maximum of 6 music therapy sessions (i.e. Music-Assisted Relaxation) during a two weeks time frame.
  Interventions: Behavioral: Music-Assisted Relaxation
- Control Group (No Intervention): Treatment as usual.

INTERVENTIONS:
Behavioral: Music-Assisted Relaxation — The music therapy sessions are based on MAR (Music-Assisted Relaxation), a music therapy technique that includes listening to live music, combined with deep diaphragmatic breathing and/or guided imagery relaxation. In a first step, the procedure will explained to the patient and he/she will be asked to close his/her eyes or focus on a fixed point on the ceiling or wall. Subsequently, a verbal introduction will be provided for fostering body and respiratory awareness. Then a mental image will be introduced (e.g., sitting on a beach watching the waves of the sea; being on top of a mountain looking at the horizon; imagining a safe and comfortable personalized place) and live music will be provided based on the principles of entrainment. The patient is asked to let himself/herself guide by the music and breath with the music while concentrating on the imagery. Once the music is over, the patient is again asked to become aware and the experience during the session will verbally discussed.
  Other Names: Music Therapy
  Arms: Intervention group

SUMMARY:
This is a randomized clinical trial studying the effectiveness of music therapy (i.e. MAR - Music-Assisted Relaxation) on pain intensity in burn patients hospitalized at the Adults Intensive Care Unit of the University Hospital Fundación Santa Fe de Bogotá in Colombia. Secondary outcome measures include anxiety and depression levels, vital signs, medication intake, quality of hospitalization and EEG, EMG, and ECG measurements. This is the first study in Colombia investigating the effectiveness of music therapy with this population.

DETAILED DESCRIPTION:
Introduction: Pain management is one of the greatest challenges in the critical care of burn patients and is frequently associated with high levels of anxiety and depression. Several studies and meta-analyses confirm the effectiveness of music interventions and music therapy in changing the experience of pain in hospitalized patients, but further clinical trials are needed investigating specific music therapy interventions in addressing pain in burn patients.

Objectives: To investigate the effect of MAR (Music-Assisted Relaxation) on the perception of pain in burn patients at the AICU (Adult Intensive Care Unit) of the Fundación Santa Fe de Bogotá (FSFB). MAR is a music therapy technique that includes listening to live music, combined with deep diaphragmatic breathing and / or guided relaxation and the use of imagery. The music applied will be based on the principles of entrainment: first, the music is synchronized with the vital signs of the patients (e.g. respiratory rate) and then musical elements (e.g. tempo) are modulated to encourage the transition to a state of deep relaxation.

Methodology: This is a randomized controlled clinical trial with an intervention group and a parallel control group. The intervention group will receive a minimum of three music therapy sessions per week up to a maximum of two weeks (6 sessions). The control group will receive treatment as usual. The main outcome measure is the intensity of perceived pain and will be measured with a Visual Analogue Scale (VAS) before and after each session. Secondary measures are: levels of anxiety and depression (HADS - Hospital Anxiety and Depression Scale); vital signs (heart rate, respiratory rate, oxygen saturation); the use of analgesic medications (complementary or rescue doses); and the quality of hospitalization perceived by the patients. Additionally, in some patients EEG (Electroencephalogram), ECG (Electrocardiography) and EMG (Electromyography) measurements will be taken, as long as the medical condition allows it. The data collection will be carried out by blinded research assistants.

Analysis: Data analysis will be carried out by a statistician from the FSFB and in collaboration with the Department of Biomedical Engineering of the Universidad de los Andes. Taking a p value of less than 5% (0.05) as clinical significance, a univariate analysis will be performed initially. Subsequently, a multivariate analysis will be performed using logistic regression to establish the contribution of each of the variables studied.

Expected results: Successful pain management is one of the most important factors in the clinical outcome of burn patients. This is the first study in Colombia that seeks to determine the effectiveness of music therapy on pain management with this population. This study will help to broaden and deepen the scientific knowledge of music therapy in the area of critical care and will promote the acquisition of new knowledge and interdisciplinary research among the institutions involved.

ELIGIBILITY:
Inclusion Criteria:

* Burn patients of legal age.
* Estimated hospitalization of > 8 days at the time of signing the informed consent.

Exclusion Criteria:

* Patients with known psychiatric disorders.
* Patients with cognitive disabilities.
* Mechanically ventilated and sedated patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | Throughout study completion, up to 2 weeks after randomization.
  Measures the change in the perceived pain intensity with a Visual Analogue Scale from 0-10 with higher scores indicating higher pain and lower scores indicating less pain.

SECONDARY OUTCOMES:
Change in anxiety and depression levels | Throughout study completion, up to 2 weeks after randomization.
  Measures changes in anxiety and depression levels with the Hospital Anxiety and Depression Scale from 0 to 21 total scores. Higher scores indicate higher levels of anxiety and depression and lower scores indicate lower levels of anxiety and depression.
Changes in heart rate | Throughout study completion, up to 2 weeks after randomization.
  Measures changes in heart rate via hospital monitors. These are changes in bpm (beats per minute) and will be averaged during a 10 minutes pre-intervention phase, during the interventions and a 10 minutes post-intervention phase.
Changes in respiratory rate | Throughout study completion, up to 2 weeks after randomization.
  Measures changes in respiratory rate via hospital monitors. These are changes in bpm (breaths per minute) and will be averaged during a 10 minutes pre-intervention phase, during the interventions and a 10 minutes post-intervention phase.
Changes in oxygen saturation | Throughout study completion, up to 2 weeks after randomization.
  Measures changes in arterial oxygen saturation (SaO2) via pulse oximetry. These are changes in percentage (%) of arterial oxygen saturation and will be averaged during a 10 minutes pre-intervention phase, during the interventions and a 10 minutes post-intervention phase.
Medication intake | Throughout study completion, up to 2 weeks after randomization.
  complementary or rescue dosis asked for by the patient
Changes in Electroencephalography | Throughout study completion, up to 2 weeks after randomization.
  Measures changes in the electrical activity of brain regions with the MicroMed 64. Measurements of the change in activity in the theta (4-8 Hz), alpha (8-12 Hz), beta 1 (12-18 Hz) and beta 2 (18-30 Hz) physiological bands will be taken from the electroencephalography records. The set up will be carried out according to international assembly 10-20, but the number of electrodes will depend on the location of the burns and the approval of the treating doctor according to each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ettenberger, PhD, Principal Investigator — Fundación Santa Fe de Bogotá
Locations (1):
- Fundación Santa Fe de Bogotá, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: Based on aims and scope of further analysis

REFERENCES:
- [Derived] Ettenberger M, Maya R, Salgado-Vasco A, Cordoba-Silva JG, Amarillo M, Betancourt-Zapata W, Marin-Sanchez J, Gomez-Ortega V, Valderrama M. The effect of music therapy on background pain, anxiety, depression, vital signs, and medication usage in adult burn patients in the Intensive Care Unit: A randomized controlled trial. Burns. 2025 Sep;51(7):107587. doi: 10.1016/j.burns.2025.107587. Epub 2025 Jun 26. PMID 40602276
- [Derived] Cordoba-Silva J, Maya R, Valderrama M, Giraldo LF, Betancourt-Zapata W, Salgado-Vasco A, Marin-Sanchez J, Gomez-Ortega V, Ettenberger M. Music therapy with adult burn patients in the intensive care unit: short-term analysis of electrophysiological signals during music-assisted relaxation. Sci Rep. 2024 Oct 9;14(1):23592. doi: 10.1038/s41598-024-73211-3. PMID 39384859
- [Derived] Ettenberger M, Maya R, Salgado-Vasco A, Monsalve-Duarte S, Betancourt-Zapata W, Suarez-Canon N, Prieto-Garces S, Marin-Sanchez J, Gomez-Ortega V, Valderrama M. The Effect of Music Therapy on Perceived Pain, Mental Health, Vital Signs, and Medication Usage of Burn Patients Hospitalized in the Intensive Care Unit: A Randomized Controlled Feasibility Study Protocol. Front Psychiatry. 2021 Oct 18;12:714209. doi: 10.3389/fpsyt.2021.714209. eCollection 2021. PMID 34733185